CLINICAL TRIAL: NCT04954547
Title: The Effect of Activities-based Subsidy on Body Fat Loss
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Noah Lim (Other)
Responsible Party: Sponsor-Investigator, Noah Lim, Professor, National University of Singapore
Organization: National University of Singapore (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: NUS-IRB-2020-643
Record Dates: First submitted 2021-06-21; First posted 2021-07-08 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Subsidy Arm (Experimental): Participants in the arm will receive $$50 if they reach the PBF goal and will be subsidized on approved health-improving expenses.
  Interventions: Behavioral: Subsidy Treatment
- Cash Arm (Experimental): Participants in the arm will receive S$350 if they reach the PBF goal.
  Interventions: Behavioral: Cash Treatment
- Control (No Intervention): Other than the participation fees, no additional incentives will be provided.

INTERVENTIONS:
Behavioral: Subsidy Treatment — Participants will be awarded $50 for reaching the PBF goal at the end of 12 weeks. Regardless of goal-attainment, participants will be reimbursed 50% of approved health-improving expenses up to a cap of $300 in the 12 weeks. The subsidy is voluntary and flexible, with no direct intervention from researchers - participants will submit receipts and simply be reimbursed at the end of the experiment (subject to approval from the research team).
  Arms: Subsidy Arm
Behavioral: Cash Treatment — Participants will be awarded $350 for reaching the PBF goal at the end of 12 weeks.
  Arms: Cash Arm

SUMMARY:
This 24-week-long study compares the effectiveness of two types of incentives for weight loss: 1) conditional subsidy 2) financial goal reward. Target participants are overweight female Singaporeans or Permanent Residents who are otherwise healthy.

DETAILED DESCRIPTION:
This study, which spans 24 weeks (12 treatment, 12 post-treatment), aims to compare the effectiveness of 2 financial incentive structures - a conditional subsidy versus a goal reward - on fat loss. 600 overweight but otherwise healthy female Singaporeans or Permanent Residents will be recruited via 2 recruitment phases, 2 months apart from each other. Participants will be given an individual-tailored percentage body fat (PBF) goal and assigned to one of three interventions:

1. Subsidy treatment group (STG) - Participants will be awarded $X for reaching the PBF goal at the end of 12 weeks. Regardless of goal attainment, participants will also be reimbursed 50% of approved health-improving expenses up to a cap of $Y in the 12 weeks. The subsidy is voluntary and flexible, with no direct intervention from researchers - participants will submit receipts to the program website and simply be reimbursed at the end of the experiment. To prevent cheating, all receipts must bear the participants' full name or be justifiably traceable to them. When submitting the receipt to the program website, they must also specify the purpose of the expense - this serves as a psychological reminder to utilize the expense more meaningfully, while allowing us to discern better to approve or reject the reimbursement claim.
2. Cash treatment group (CTG). Participants will be awarded $(X+Y) for reaching the PBF goal at the end of 12 weeks.
3. Control. Other than the participation fees, no additional incentives will be provided.

All participants will be given an individual-tailored 12-week PBF goal. The formula for this goal will be set following the approval of the IRB, in consultation with medical and fitness professionals (including certified doctors and fitness trainers) to ensure that it is safe, challenging, and achievable. The base formula, which assumes a 5% weight loss as is often defined to be the medically significant level, is:

(P*W-x*5%*W)/(95%*W)

where P is PBF at baseline (week 1), W is body mass in kg at baseline, P×W is their body fat mass at baseline, and x, ranging between 0% and 100%, is the parameter that is set in consultation with professionals. At 100%, it implies that all 5% in weight loss is from fat, vice versa.

Because P and W differ between most persons, our formula tailors a different goal to each research subject. Our formula is meant to be flexible toward each participant's baseline weight and body fat percent. Leveraging the 5% weight loss target, the investigators determined the expected percentage of this weight that is lost as fat, knowing that weight loss includes not only fat loss but also other components such as water loss. In previous studies, for 1 kg loss in weight, on average, 78.8% came from body fat. Hence, the investigators have targeted 80% of weight loss from our participants to come from body fat.

To examine changes in health, objective measurements will be made during scheduled participant visits on Weeks 1, 12, and 24. Measures include height, weight, waist circumference, and PBF. Each participant will also be given a free digital scale for personal use from home. Their weight and PBF data from the scale will be synchronized to a mobile application, which we will retrieve with the participant's consent, to examine changes throughout the study's duration.

There are a total of 3 scheduled visits. The first in Week 1 allows us to determine the baseline measures. The second visit in Week 12 marks the end of the treatment and allows us to investigate treatment effects. The last visit in Week 24 checks for post-treatment effects. During all 3 visits, the participants will also complete a Health Risk Assessment Survey. This survey should take no longer than 10 minutes to complete, and the research team will be physically present to assist them with it if so required.

Due to the uncertainty of the pandemic, the investigators may hold the second and/or the third research visits virtually (or at least provide an online option) to avoid large gatherings if necessary. For each virtual research visit, the research team will contact the participants through a video call, during which they will step on the weighing scales and show the readings to the team. If a research visit is held online, the participation fee/rewards will be sent electronically. The research team will still hold physical meetings for those who experience technical difficulties.

To let participants track their PBF progress, every participant would be given a digital scale for their keeping even after the research has concluded. The scale, named 'Lite Mould Body Composition Smart Scale', priced at US$13 (before shipping) is commercially available and will be supplied by the manufacturer 'Yolanda'. It comes with a free mobile application to let them track their progress. The app is publicly available on the Apple and Google Play stores for free under the name 'Feelfit' by Shenzhen QingNiu Software Co. Ltd. Referring to the Health Products Act (HPA), this scale would not be defined as a "medical device". The digital scale serves simply, as would a conventional scale, to inform the user on some bodily metric. It does not attempt to make any medical judgment or recommendation for the user. The research team has done testing on the digital scale and is satisfied with the precision of the device. The participants are expected to weigh-in on the scales weekly from home at their convenience. In the middle of each of the 12 weeks (e.g. Wednesday or Thursday), an automated email will be sent to the participants reminding them to do so by the end of the week (Sunday). Non-compliance will not be penalized, but participants are strongly encouraged to weigh-in. The following is the complete list of data that the participants will have access to from the scale's mobile application. The researchers, with the participants' consent, will also retrieve this data for analysis: 1. Basal metabolism rate; 2. BMI; 3. Bone mass; 4. Metabolic age; 5. Muscle mass; 6. PBF; 7. Skeletal muscle weight ratio; 8. Subcutaneous fat; 9. Total body water; 10. Visceral fat; 11. Weight

The study will be split into two waves of 300 participants. The investigators will start the first wave when they successfully recruit 300 eligible participants in the first recruitment phase and the second wave with another 300 eligible participants in the second recruitment phase.

ELIGIBILITY:
Inclusion Criteria:

* Singaporeans or Permanent Residents
* Female
* Overweight (BMI: 23 to 27.5)
* Participants need to own a smartphone or tablet
* Must be able to commit to a 24-week research program focused on improving health
* Own a smartphone or tablet

Exclusion Criteria:

* Chronically diseased (e.g. hypertension, hyperglycemia, hyperlipidemia), or is suffering or suffered from medical conditions (e.g. stroke, heart attack).
* Currently pregnant or breastfeeding or intending to become pregnant over the next year
* Currently participating in any other research program focused on physical activity or weight loss
* Currently taking any prescribed medications.

Ages: 25 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 800 (Estimated)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Whether reaching the prescribed PBF goal | At the end of the 12 weeks
  This is binary variable, which is 1 if the participant reaches the prescribed PBF goal, and 0 otherwise
Whether maintaining what has achieved in the post-treatment period | At the end of the 24 weeks
  This is binary variable, which is 1 if the participant loses more fat in the post-treatment period than in the intervention period, and 0 otherwise.
Achievement Percentage | At the end of the 24 weeks
  A percentage of the change in PBF from the predetermined change in PBF
Weekly Achievement Percentage | Through study completion (24 weeks)
  A percentage of the change in PBF from the predetermined change in PBF

CONTACTS AND LOCATIONS:
Overall Officials: Noah Lim, PhD, Study Director — The Global Asia Institute, The National University of Singapore; Andrea Chung, PhD, Principal Investigator — Booz Allen Hamilton; Ta-Cheng Huang, PhD, Principal Investigator — The Global Asia Institute, The National University of Singapore; Kegon Tan, PhD, Principal Investigator — University of Rochester
Locations (1):
- National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chaston TB, Dixon JB, O'Brien PE. Changes in fat-free mass during significant weight loss: a systematic review. Int J Obes (Lond). 2007 May;31(5):743-50. doi: 10.1038/sj.ijo.0803483. Epub 2006 Oct 31. PMID 17075583